CLINICAL TRIAL: NCT06058208
Title: The Effect of Baby Smell and Visual Stimulus Program on Mothers' Cortical and Breast Oxygenation, Milk Amount and Mother-Infant Attachment: Randomized Controlled Study
Brief Title: Baby Smell Visual Stimulus Program Cortical and Breast Oxygenation Milk Amount Mother-Infant Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Proffessor Doktor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUnı4244
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Delivery Affecting Fetus; Preterm Labor
Keywords: breastmilk; cortical and breast oxygenation; infant odor; mother-infant bonding; NIRS; visual stimulus
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Photic Stimulation

STUDY DESIGN:
Intervention Model Description: In this randomized controlled study, "block randomization" method, which is one of the "fixed probability randomization" methods, was used in randomization. Each of the experimental and control groups was represented by one of the letters A, B, C. In the creation of the 6-block (2A, 2B, 2C) design for 54 samples and three groups; Using the "permutation" method, the assignment of 9 blocks out of 90 block options was carried out through the random numbers table on the www.random.org site. Which of the experimental and control groups will match the letters A, B, C; It was determined by the lottery method drawn by hand by the independent clinical nurse from the study. As a result of the draw, A: smell, B: smell + video, C: represented the control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baby Smell Group (Experimental): Firstly the baby beret worn by the researcher on the baby will be removed at the end of the 12th hour (at the 12th hour and 24th hour of the hospitalization in the clinic) and taken to the Obstetrics and Gynecology Service on the same floor as the NICU without waiting;Odor stimulation will be applied in the form of 30 sec odor-30 sec standby-30 sec odor-30 sec standby-30 sec odor. A total of 4 rSO2 values, including the initial value and the average of the values during three 30 sec stimulation, will be recorded in the "Cortical and Breast Oxygenation Follow-up Form". The amount of the first amount of milk, the total amount of milk until the 12th hour, the amount of oral fluid intake, the amount of milk until the 24th hour (12th hour -24th hour) and the amount of oral fluid intake will be recorded in the Milk Amount Follow-up Form.
  Interventions: Behavioral: Olfactory stimulation
- Baby Smell and Visual Stimulus Group (Experimental): Firstly the baby video (visual stimulus) and beret worn by the researcher on the baby will be removed at the end of the 12th hour (at the 12th hour and 24th hour of the hospitalization in the clinic) taken by researcher and taken to the clinic on the same floor as the NICU without waiting; Once the initial rSO2 value has been recorded, the mother will be instructed to sniff the beret uninterruptedly until further warning by the researcher and to watch the image of her baby unfolding on the tablet fixed to the floor during the entire measurement process. Odor stimulation to the mother will be applied in the form of 30 sec odor-30 sec waiting-30 sec odor-30 sec waiting-30 sec odor respectively, and visual stimulation will be applied as uninterrupted 2.5 min. At the end of 24 hours, the Mother-Baby Interaction Form and the MIBS tool will be re-applied as the final test.
  Interventions: Behavioral: Olfactory stimulation; Behavioral: Visual stimulation
- Control Group (No Intervention): The intervention and data collection process in the control group is the same as the intervention in the odor group; As a placebo instead of odor stimulation, the odorless beret will be offered in the same conditions.

INTERVENTIONS:
Behavioral: Olfactory stimulation — Olfactory stimulation: Mothers will be made to smell their babies' odor.
  Arms: Baby Smell Group; Baby Smell and Visual Stimulus Group
Behavioral: Visual stimulation — Mothers will be shown video images of their babies.
  Arms: Baby Smell and Visual Stimulus Group

SUMMARY:
In this study, the effect of infant odor and visual stimulus program applied to mothers who had delivered by cesarean section and whose babies were taken to the NICU on cortical and breast oxygenation (rSO2), amount of breast milk and mother-infant bonding was investigated.

DETAILED DESCRIPTION:
One of the conditions that prevent the preterm baby from being close to the mother in the early period is cesarean delivery and subsequent removal to the NICU. In the first hour of life, the process immediately after birth, when the newborn is alert, makes eye contact, focuses, finds the unaided mother's breast and begins to feed, deteriorates in babies in need of intensive care and mothers begin the experience of parenting with delayed attachment. The mother experiences high levels of stress due to changes in many parental roles such as being physically separated from her baby, not being able to breastfeed effectively, not being able to care for her baby and the intensive care environment, and experiencing a delay in lactation with the effect of cesarean delivery. In the literature, many interventions have been implemented to reduce the negative effects of mother-infant separation on lactation and attachment in mothers who have given birth by cesarean section. However, there is no published research examining the effect of infant odor and visual stimulus program applied to mothers who had delivered by cesarean section and whose babies were taken to the NICU on cortical and breast oxygenation (rSO2), amount of breast milk and mother-infant bonding. In addition, being able to assess how the mother's cortical and breast oxygenation changes while smelling her baby's scent and watching her/his video will further strengthen the results of the measurement tools.

ELIGIBILITY:
Inclusion Criteria:

Infant

* Born at 28-37 (36+6) weeks of gestation
* Admission to the NICU in the same hospital as the mother immediately after birth Mother
* To agree to participate in the study,
* To give birth by cesarean section,
* To be able to use the Turkish language,
* To pass the smell test (to correctly identify the 3 different types of smell presented),
* Not to have been diagnosed with depression etc. Psychiatry at the time of the study

Exclusion Criteria:

Infant

* The presence of conditions that affect the baby's original smell (baby born with Meconium, Hepatitis C and HIV infected baby)
* Infant who underwent interventional intervention in the head area
* The baby whose suction function is sufficient and who can suck breast milk

Mother

* Admission to Intensive Care,
* Being covid positive (as the sense of smell will be affected),
* Having a mental, neurological, nasal related disease,
* Having a communication problem

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Cortical and Breast Oxygenation Follow-up Parameter | First measurement- At 12th hour of the postpartum period.
  Form; was created by the researcher in accordance with the literature to record cortical and breast oxygenation (Tanimoto et al., 2011; Schafer et al., 2019). NIRS measurement range was accepted as 15-95 for breast and cortical oxygenation. In the study of Tanimoto et al. (2011), the average of the measurement periods of 30 seconds was taken as the initial value; A 5-minute chart has been generated. Similarly in our study; The initial rSO2 value for both cortical and breast will be recorded, and the average rSO2 value for each block will be recorded during 30 seconds of intervention (smell, odor + visual stimulus, control) repeated 3 times. The form contains two charts with 4 cortical and breast rSO2 recordings for the measurement to be made at two different times (12th and 24th hour of birth)
Cortical and Breast Oxygenation Follow-up Parameter | Second measurement- At 24th hour of the postpartum period.
  Form; was created by the researcher in accordance with the literature to record cortical and breast oxygenation (Tanimoto et al., 2011; Schafer et al., 2019). NIRS measurement range was accepted as 15-95 for breast and cortical oxygenation. In the study of Tanimoto et al. (2011), the average of the measurement periods of 30 seconds was taken as the initial value; A 5-minute chart has been generated. Similarly in our study; The initial rSO2 value for both cortical and breast will be recorded, and the average rSO2 value for each block will be recorded during 30 seconds of intervention (smell, odor + visual stimulus, control) repeated 3 times. The form contains two charts with 4 cortical and breast rSO2 recordings for the measurement to be made at two different times (12th and 24th hour of birth)
Milk Amount Follow-up Form | First measurement- At 12th hour of the postpartum period.
  It was created by the researcher in line with the literature (Turhan, 2020). The form will record the amount of initial milking, the total amount of milk up to the 12th hour, and the amount of oral fluid intake, the total amount of milk between the 12th-24th hour onwards, and the amount of oral fluid intake.
Milk Amount Follow-up Form | Second measurement- At 24th hour of the postpartum period.
  It was created by the researcher in line with the literature (Turhan, 2020). The form will record the amount of initial milking, the total amount of milk up to the 12th hour, and the amount of oral fluid intake, the total amount of milk between the 12th-24th hour onwards, and the amount of oral fluid intake.
Mother to Infant Bonding Scale | First measurement- Within 1 hour of the postpartum period.
  The "Mother to Infant Bonding Scale" tool developed by Taylor et al., (2005) was adapted into Turkish by Karakulak Aydemir and Alparslan, (2016). The scale, which is arranged in such a way that it can be applied from the first day after birth and allows the mother to express her feelings towards her baby with a single word, consists of 8 items and is in the form of 4 likerts. The score range of the scale is between 0-24. A high score indicates low bonding.
Mother to Infant Bonding Scale | Second measurement- At 24th hour of the postpartum period.
  The "Mother to Infant Bonding Scale" tool developed by Taylor et al., (2005) was adapted into Turkish by Karakulak Aydemir and Alparslan, (2016). The scale, which is arranged in such a way that it can be applied from the first day after birth and allows the mother to express her feelings towards her baby with a single word, consists of 8 items and is in the form of 4 likerts. The score range of the scale is between 0-24. A high score indicates low bonding.
Mother and Infant Information Tool | First measurement- Within 1 hour of the postpartum period.
  According to the literature (Tanimoto et al., 2011; Croy et al., 2019; Schafer et al., 2020) consists of questions compiled by the researcher including the demographic characteristics of the mother (age, educational status) obstetric and clinical characteristics (pregnancy planning status, anesthesia method), characteristics of the baby (gender, gestational week, birth weight, medical diagnosis, nutrition type).

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Küçükoğlu, Prof, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Croy I, Frackowiak T, Hummel T, Sorokowska A. Babies Smell Wonderful to Their Parents, Teenagers Do Not: an Exploratory Questionnaire Study on Children's Age and Personal Odor Ratings in a Polish Sample. Chemosens Percept. 2017;10(3):81-87. doi: 10.1007/s12078-017-9230-x. Epub 2017 Jun 27. PMID 28932343
- [Background] Durkaya Göktepe, G., 2021. "Maternal infant bonding and affecting factors in the early period in women who have term and preterm birth" Unpublished Master's Thesis, Istanbul University-Cerrahpaşa Graduate Education Institute, Istanbul
- [Background] Karakulak, H.A., Alparslan, Ö., 2016. "Adaptation of Mother to Infant Bonding Scale to The Turkish Society: Aydın Sample", Çağdaş Journal of Medicine, 6(3), 188-199.
- [Background] Schafer L, Hummel T, Croy I. The Design Matters: How to Detect Neural Correlates of Baby Body Odors. Front Neurol. 2019 Jan 16;9:1182. doi: 10.3389/fneur.2018.01182. eCollection 2018. PMID 30700979
- [Background] Schafer L, Sorokowska A, Sauter J, Schmidt AH, Croy I. Body odours as a chemosignal in the mother-child relationship: new insights based on an human leucocyte antigen-genotyped family cohort. Philos Trans R Soc Lond B Biol Sci. 2020 Jun 8;375(1800):20190266. doi: 10.1098/rstb.2019.0266. Epub 2020 Apr 20. PMID 32306871
- [Background] Tanimoto K, Kusaka T, Nishida T, Ogawa K, Kato I, Ijichi S, Mikami J, Sobue I, Isobe K, Itoh S. Hemodynamic changes in the breast and frontal cortex of mothers during breastfeeding. Pediatr Res. 2011 Oct;70(4):400-5. doi: 10.1203/PDR.0b013e31822a363a. PMID 21705961
- [Background] Taylor A, Atkins R, Kumar R, Adams D, Glover V. A new Mother-to-Infant Bonding Scale: links with early maternal mood. Arch Womens Ment Health. 2005 May;8(1):45-51. doi: 10.1007/s00737-005-0074-z. Epub 2005 May 4. PMID 15868385
- [Background] Turhan, İ., 2020. "The effect of monitoring the video image of the baby on the mother's milk and maternal connectivity to the mother in the newborn unit of the infant" (Unpublished Master's Thesis), Erciyes University/ Institute of Health Sciences, Kayseri.